CLINICAL TRIAL: NCT05779111
Title: A Retrospective Analysis: Whether Five Factors Affect PFS in Patients With Locally Advanced Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CQGOG0111
Record Dates: First submitted 2023-02-19; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Locally Advanced Cervical Cancer; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scores greater than or equal to 3 in patients with locally advanced cervical cancer: Scores greater than or equal to 3 in patients with locally advanced cervical cancer
- Patients with locally advanced cervical cancer scored less than 3 points: Patients receiving radiotherapy for locally advanced cervical cancer were scored according to five factors, with a score of less than 3

SUMMARY:
In previous studies, the investigators found that five factors were effective in predicting the probability of locally advanced cervical cancer with para-aortic lymph node metastasis.A retrospective study was conducted to explore the influence of 5 factors on PFS in patients with locally advanced cervical cancer receiving radiotherapy and chemotherapy.

DETAILED DESCRIPTION:
In previous studies, the investigators found that five factors were effective in predicting the probability of locally advanced cervical cancer with para-aortic lymph node metastasis.5 factors included positive iliac lymph nodes, histological type, tumor size, positive pelvic lymph nodes on both sides, and maximum lymph node diameter greater than 1cm. Different factors give different scores.If the score is higher than 3, the probability of retroperitoneal lymph node metastasis in patients with locally advanced cervical cancer is significantly increased, and the prognosis of patients is affected. Patients with locally advanced cervix receiving radical radiotherapy were scored based on 5 factors.Patients with scores greater than or equal to 3 points were compared with patients with scores less than 3 points.

ELIGIBILITY:
Locally advanced cervical cancer patients receiving radiotherapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From May 2016 to July 2021, 183 patients with locally advanced cervical cancer received radiotherapy in our hospital ,with or without chemotherapy.Patients were scored according to 5 factors. PFS were compared between patients with scores greater than or equal to 3 points and those with scores less than 3 points. PFS is defined as the time from the end of treatment to disease progression or the time of the last follow-up 2022-10-01.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival（PFS） | 3 months
  Whether there are differences in PFS between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Zou Dongling, M.D., Study Director — Chongqing University Cancer Hospital Chongqing, Chongqing, China,
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No